CLINICAL TRIAL: NCT04696120
Title: Effects of APIXaban on BRAIN Protection in Patients With Sinus Rhythm and Heart Failure: APIXBRAIN-HF Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Dt&Sanomedics (Industry)
Responsible Party: Principal Investigator, Eung Ju Kim, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020GR0592
Record Dates: First submitted 2021-01-03; First posted 2021-01-06 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure; Sinus Rhythm; Cerebrovascular Disease
Keywords: Heart failure; Sinus rhythm; NOAC; Brain
MeSH Terms: conditions — Heart Failure; Cerebrovascular Disorders | interventions — apixaban; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group: apixaban (Experimental): apixaban 2.5mg or 5mg bid
  Interventions: Drug: Apixaban
- Control group: placebo (Placebo Comparator): placebo bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban — Patients who are randomly assigned to apixaban group will receive apixaban 5mg or 2.5mg bid
  Other Names: apixaban 5mg or 2.5mg bid
  Arms: Study group: apixaban
Drug: Placebo — All patients who are assigned to placebo group will receive placebo
  Other Names: placebo bid
  Arms: Control group: placebo

SUMMARY:
objectives: The primary aim of APIXBRAIN-HF Trial is to explore the effects of apixaban on brain protection in patients with sinus rhythm and heart failure

Primary / Secondary Endpoint

1. New occurrence of brain pathology 1) Cortical cerebral microinfarcts 2) Silent lacunar infarction 3)Progression of white matter hyperintensities
2. Secondary endpoint 1) The change of cognitive function evaluated by MMSE-2 2) Individual variable of primary endpoint
3. Safety Endpoint Evaluation 1) Cerebral microbleeds on imaging

DETAILED DESCRIPTION:
This study is a double-blind, parallel-group, and randomization study. The investigators will enroll the patients with heart failure who demonstrated LV systolic dysfunction (LVEF ≤ 40%) and sinus rhythm with a CHA2DS2-VASc score ≥ 3. All patients would be randomly assigned to either the apixaban group or placebo group. Patients assigned to the apixaban group will receive 5mg bid or 2.5mg bid (patients with at least 2 of the following characteristics: aged≥80-year, bodyweight ≤60kg, serum creatinine 1.5 ml/dL) and patients in the placebo group will receive a placebo of apixaban. Both drugs will be maintained for 6 months. During the study period, all patients will be carefully monitored for thromboembolic events, including stroke. At the beginning of the study and 6 months after randomization, 3T Brain MRI and MMSE-2 test will be performed to identify changes in brain structure and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 19 years old
* Patients with sinus rhythm
* Newly diagnosed of heart failure or aggravated heart failure symptom

  1. Dyspnea (≥ NYHA II)
  2. plasma BNP ≥ 200 pg/ml or NT-proBNP ≥ 800 pg/ml
* LV systolic dysfunction on echocardiography within 3 month of enrollment

  1) LVEF ≤ 40%
* Those with CHA2DS2-VASc ≥ 3
* Modified Rankin Score ≤ 4

Exclusion Criteria:

* Patients already subscribed warfarin or antiplatelet therapy or have clear indication for warfarin or antiplatelet therapy
* At high risk for bleeding
* Patients with atrial fibrillation
* Estimated glomerular filtration rate (CKD-EPI formula) < 15 ml/min/1.73 m2)
* Recent stroke or brain hemorrhage (within 3 months)
* Patients who was diagnosed of myocardial infarction or who has plan to PCI/CABG at enrollment
* End stage heart failure with life expectancy ≤ 6 months
* Patients with bed ridden status (Modified Rankin Score ≥ 5)
* Patients with liver dysfunction (AST, ALT > 2 times of upper normal limits or total bilirubin > 1.5 of upper normal limits)
* At of pregnancy or breastfeeding
* Patients who disagree with the use of medically acceptable contraception during the clinical trial period
* Patients with contraindication of apixaban

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-02 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
New occurrence of brain pathology | 24 weeks
  1) Cortical cerebral microinfarcts 2) Silent lacunar infarction 3)Progression of white matter hyperintensities

SECONDARY OUTCOMES:
The change of Mini-Mental State Examination-2 (MMSE-2) score | 24 weeks
  The change of Mini-Mental State Examination-2 (MMSE-2) score compared to baseline. Higher scores mean a better outcome.
New occurrence of cortical cerebral microinfarcts | 24 weeks
  New occurrence of cortical cerebral microinfarcts compared to baseline
New occurrence of silent lacunar infarction | 24 weeks
  New occurrence of silent lacunar infarction compared to baseline
Progression of white matter hyperintensities (more than 10% increase) | 24 weeks
  Progression of white matter hyperintensities (more than 10% increase) compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eung Ju Kim, MD, PhD., Principal Investigator — Professor
Locations (10):
- South Korea (10):
  - Korea University Guro Hospital, Seoul, Guro-gu
  - Korea University Ansan Hospital, Ansan
  - Chungnam National University Hospital, Daejeon
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Anker SD, AlHabib KF, Cowie MR, Force TL, Hu S, Jaarsma T, Krum H, Rastogi V, Rohde LE, Samal UC, Shimokawa H, Budi Siswanto B, Sliwa K, Filippatos G. Heart failure: preventing disease and death worldwide. ESC Heart Fail. 2014 Sep;1(1):4-25. doi: 10.1002/ehf2.12005. PMID 28834669
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990
- [Background] Nichols GA, Reynolds K, Kimes TM, Rosales AG, Chan WW. Comparison of Risk of Re-hospitalization, All-Cause Mortality, and Medical Care Resource Utilization in Patients With Heart Failure and Preserved Versus Reduced Ejection Fraction. Am J Cardiol. 2015 Oct 1;116(7):1088-92. doi: 10.1016/j.amjcard.2015.07.018. Epub 2015 Jul 15. PMID 26235928
- [Background] Maggioni AP, Dahlstrom U, Filippatos G, Chioncel O, Crespo Leiro M, Drozdz J, Fruhwald F, Gullestad L, Logeart D, Fabbri G, Urso R, Metra M, Parissis J, Persson H, Ponikowski P, Rauchhaus M, Voors AA, Nielsen OW, Zannad F, Tavazzi L; Heart Failure Association of the European Society of Cardiology (HFA). EURObservational Research Programme: regional differences and 1-year follow-up results of the Heart Failure Pilot Survey (ESC-HF Pilot). Eur J Heart Fail. 2013 Jul;15(7):808-17. doi: 10.1093/eurjhf/hft050. Epub 2013 Mar 28. PMID 23537547
- [Background] Ziaeian B, Fonarow GC. Epidemiology and aetiology of heart failure. Nat Rev Cardiol. 2016 Jun;13(6):368-78. doi: 10.1038/nrcardio.2016.25. Epub 2016 Mar 3. PMID 26935038
- [Background] Mamas MA, Sperrin M, Watson MC, Coutts A, Wilde K, Burton C, Kadam UT, Kwok CS, Clark AB, Murchie P, Buchan I, Hannaford PC, Myint PK. Do patients have worse outcomes in heart failure than in cancer? A primary care-based cohort study with 10-year follow-up in Scotland. Eur J Heart Fail. 2017 Sep;19(9):1095-1104. doi: 10.1002/ejhf.822. Epub 2017 May 3. PMID 28470962
- [Background] Kim W, Kim EJ. Heart Failure as a Risk Factor for Stroke. J Stroke. 2018 Jan;20(1):33-45. doi: 10.5853/jos.2017.02810. Epub 2018 Jan 31. PMID 29402070
- [Background] Divani AA, Vazquez G, Asadollahi M, Qureshi AI, Pullicino P. Nationwide frequency and association of heart failure on stroke outcomes in the United States. J Card Fail. 2009 Feb;15(1):11-6. doi: 10.1016/j.cardfail.2008.09.001. Epub 2008 Dec 25. PMID 19181288
- [Background] Hays AG, Sacco RL, Rundek T, Sciacca RR, Jin Z, Liu R, Homma S, Di Tullio MR. Left ventricular systolic dysfunction and the risk of ischemic stroke in a multiethnic population. Stroke. 2006 Jul;37(7):1715-9. doi: 10.1161/01.STR.0000227121.34717.40. Epub 2006 Jun 1. PMID 16741172
- [Background] Pullicino P, Homma S. Stroke in heart failure: atrial fibrillation revisited? J Stroke Cerebrovasc Dis. 2010 Jan;19(1):1-2. doi: 10.1016/j.jstrokecerebrovasdis.2009.09.002. No abstract available. PMID 20123219
- [Background] Haeusler KG, Laufs U, Endres M. Chronic heart failure and ischemic stroke. Stroke. 2011 Oct;42(10):2977-82. doi: 10.1161/STROKEAHA.111.628479. Epub 2011 Sep 8. PMID 21903953
- [Background] Adelborg K, Szepligeti S, Sundboll J, Horvath-Puho E, Henderson VW, Ording A, Pedersen L, Sorensen HT. Risk of Stroke in Patients With Heart Failure: A Population-Based 30-Year Cohort Study. Stroke. 2017 May;48(5):1161-1168. doi: 10.1161/STROKEAHA.116.016022. Epub 2017 Apr 4. PMID 28377383
- [Background] Kang SH, Kim J, Park JJ, Oh IY, Yoon CH, Kim HJ, Kim K, Choi DJ. Risk of stroke in congestive heart failure with and without atrial fibrillation. Int J Cardiol. 2017 Dec 1;248:182-187. doi: 10.1016/j.ijcard.2017.07.056. Epub 2017 Jul 20. PMID 28826798
- [Background] Abdul-Rahim AH, Perez AC, MacIsaac RL, Jhund PS, Claggett BL, Carson PE, Komajda M, McKelvie RS, Zile MR, Swedberg K, Yusuf S, Pfeffer MA, Solomon SD, Lip GYH, Lees KR, McMurray JJV; Candesartan in Heart failure Assessment of Reduction in Mortality and Morbidity-Preserved (CHARM-Preserved) and the Irbesartan in Heart Failure with Preserved Systolic Function (I-Preserve) Steering Committees. Risk of stroke in chronic heart failure patients with preserved ejection fraction, but without atrial fibrillation: analysis of the CHARM-Preserved and I-Preserve trials. Eur Heart J. 2017 Mar 7;38(10):742-750. doi: 10.1093/eurheartj/ehw509. PMID 28426886
- [Background] Abdul-Rahim AH, Perez AC, Fulton RL, Jhund PS, Latini R, Tognoni G, Wikstrand J, Kjekshus J, Lip GY, Maggioni AP, Tavazzi L, Lees KR, McMurray JJ; Investigators of the Controlled Rosuvastatin Multinational Study in Heart Failure (CORONA); GISSI-Heart Failure (GISSI-HF) Committees and Investigators. Risk of Stroke in Chronic Heart Failure Patients Without Atrial Fibrillation: Analysis of the Controlled Rosuvastatin in Multinational Trial Heart Failure (CORONA) and the Gruppo Italiano per lo Studio della Sopravvivenza nell'Insufficienza Cardiaca-Heart Failure (GISSI-HF) Trials. Circulation. 2015 Apr 28;131(17):1486-94; discussion 1494. doi: 10.1161/CIRCULATIONAHA.114.013760. Epub 2015 Mar 25. PMID 25810334
- [Background] Kalaria VG, Passannante MR, Shah T, Modi K, Weisse AB. Effect of mitral regurgitation on left ventricular thrombus formation in dilated cardiomyopathy. Am Heart J. 1998 Feb;135(2 Pt 1):215-20. doi: 10.1016/s0002-8703(98)70084-5. PMID 9489967
- [Background] Lip GY, Gibbs CR. Does heart failure confer a hypercoagulable state? Virchow's triad revisited. J Am Coll Cardiol. 1999 Apr;33(5):1424-6. doi: 10.1016/s0735-1097(99)00033-9. PMID 10193748
- [Background] Vogels RL, van der Flier WM, van Harten B, Gouw AA, Scheltens P, Schroeder-Tanka JM, Weinstein HC. Brain magnetic resonance imaging abnormalities in patients with heart failure. Eur J Heart Fail. 2007 Oct;9(10):1003-9. doi: 10.1016/j.ejheart.2007.07.006. Epub 2007 Aug 23. PMID 17719270
- [Background] Havakuk O, King KS, Grazette L, Yoon AJ, Fong M, Bregman N, Elkayam U, Kloner RA. Heart Failure-Induced Brain Injury. J Am Coll Cardiol. 2017 Mar 28;69(12):1609-1616. doi: 10.1016/j.jacc.2017.01.022. PMID 28335844
- [Background] Frey A, Sell R, Homola GA, Malsch C, Kraft P, Gunreben I, Morbach C, Alkonyi B, Schmid E, Colonna I, Hofer E, Mullges W, Ertl G, Heuschmann P, Solymosi L, Schmidt R, Stork S, Stoll G. Cognitive Deficits and Related Brain Lesions in Patients With Chronic Heart Failure. JACC Heart Fail. 2018 Jul;6(7):583-592. doi: 10.1016/j.jchf.2018.03.010. Epub 2018 Jun 6. PMID 29885954
- [Background] Homma S, Thompson JL, Pullicino PM, Levin B, Freudenberger RS, Teerlink JR, Ammon SE, Graham S, Sacco RL, Mann DL, Mohr JP, Massie BM, Labovitz AJ, Anker SD, Lok DJ, Ponikowski P, Estol CJ, Lip GY, Di Tullio MR, Sanford AR, Mejia V, Gabriel AP, del Valle ML, Buchsbaum R; WARCEF Investigators. Warfarin and aspirin in patients with heart failure and sinus rhythm. N Engl J Med. 2012 May 17;366(20):1859-69. doi: 10.1056/NEJMoa1202299. Epub 2012 May 2. PMID 22551105
- [Background] Cokkinos DV, Haralabopoulos GC, Kostis JB, Toutouzas PK; HELAS investigators. Efficacy of antithrombotic therapy in chronic heart failure: the HELAS study. Eur J Heart Fail. 2006 Jun;8(4):428-32. doi: 10.1016/j.ejheart.2006.02.012. Epub 2006 Jun 5. PMID 16737850
- [Background] Cleland JG, Findlay I, Jafri S, Sutton G, Falk R, Bulpitt C, Prentice C, Ford I, Trainer A, Poole-Wilson PA. The Warfarin/Aspirin Study in Heart failure (WASH): a randomized trial comparing antithrombotic strategies for patients with heart failure. Am Heart J. 2004 Jul;148(1):157-64. doi: 10.1016/j.ahj.2004.03.010. PMID 15215806
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. Circulation. 2017 Aug 8;136(6):e137-e161. doi: 10.1161/CIR.0000000000000509. Epub 2017 Apr 28. No abstract available. PMID 28455343
- [Background] Corrigendum to: 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2018 Apr 1;39(13):1109. doi: 10.1093/eurheartj/ehx039. No abstract available. PMID 28369313
- [Background] Greenberg B, Neaton JD, Anker SD, Byra WM, Cleland JGF, Deng H, Fu M, La Police DA, Lam CSP, Mehra MR, Nessel CC, Spiro TE, van Veldhuisen DJ, Vanden Boom CM, Zannad F. Association of Rivaroxaban With Thromboembolic Events in Patients With Heart Failure, Coronary Disease, and Sinus Rhythm: A Post Hoc Analysis of the COMMANDER HF Trial. JAMA Cardiol. 2019 Jun 1;4(6):515-523. doi: 10.1001/jamacardio.2019.1049. PMID 31017637
- [Background] Zannad F, Anker SD, Byra WM, Cleland JGF, Fu M, Gheorghiade M, Lam CSP, Mehra MR, Neaton JD, Nessel CC, Spiro TE, van Veldhuisen DJ, Greenberg B; COMMANDER HF Investigators. Rivaroxaban in Patients with Heart Failure, Sinus Rhythm, and Coronary Disease. N Engl J Med. 2018 Oct 4;379(14):1332-1342. doi: 10.1056/NEJMoa1808848. Epub 2018 Aug 27. PMID 30146935
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Noseworthy PA, Yao X, Abraham NS, Sangaralingham LR, McBane RD, Shah ND. Direct Comparison of Dabigatran, Rivaroxaban, and Apixaban for Effectiveness and Safety in Nonvalvular Atrial Fibrillation. Chest. 2016 Dec;150(6):1302-1312. doi: 10.1016/j.chest.2016.07.013. Epub 2016 Sep 28. PMID 27938741
- [Background] Melgaard L, Gorst-Rasmussen A, Lane DA, Rasmussen LH, Larsen TB, Lip GY. Assessment of the CHA2DS2-VASc Score in Predicting Ischemic Stroke, Thromboembolism, and Death in Patients With Heart Failure With and Without Atrial Fibrillation. JAMA. 2015 Sep 8;314(10):1030-8. doi: 10.1001/jama.2015.10725. PMID 26318604
- [Background] Mehra MR, Vaduganathan M, Fu M, Ferreira JP, Anker SD, Cleland JGF, Lam CSP, van Veldhuisen DJ, Byra WM, Spiro TE, Deng H, Zannad F, Greenberg B. A comprehensive analysis of the effects of rivaroxaban on stroke or transient ischaemic attack in patients with heart failure, coronary artery disease, and sinus rhythm: the COMMANDER HF trial. Eur Heart J. 2019 Nov 21;40(44):3593-3602. doi: 10.1093/eurheartj/ehz427. PMID 31461239
- [Background] Lip GY, Rasmussen LH, Skjoth F, Overvad K, Larsen TB. Stroke and mortality in patients with incident heart failure: the Diet, Cancer and Health (DCH) cohort study. BMJ Open. 2012 Jul 7;2(4):e000975. doi: 10.1136/bmjopen-2012-000975. Print 2012. PMID 22773537
- [Background] Alberts VP, Bos MJ, Koudstaal P, Hofman A, Witteman JC, Stricker B, Breteler M. Heart failure and the risk of stroke: the Rotterdam Study. Eur J Epidemiol. 2010 Nov;25(11):807-12. doi: 10.1007/s10654-010-9520-y. PMID 21061046
- [Background] Witt BJ, Brown RD Jr, Jacobsen SJ, Weston SA, Ballman KV, Meverden RA, Roger VL. Ischemic stroke after heart failure: a community-based study. Am Heart J. 2006 Jul;152(1):102-9. doi: 10.1016/j.ahj.2005.10.018. PMID 16824838
- [Background] Hassell ME, Nijveldt R, Roos YB, Majoie CB, Hamon M, Piek JJ, Delewi R. Silent cerebral infarcts associated with cardiac disease and procedures. Nat Rev Cardiol. 2013 Dec;10(12):696-706. doi: 10.1038/nrcardio.2013.162. Epub 2013 Oct 29. PMID 24165909
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Jansson M, Sjalander S, Sjogren V, Renlund H, Norrving B, Sjalander A. Direct comparisons of effectiveness and safety of treatment with Apixaban, Dabigatran and Rivaroxaban in atrial fibrillation. Thromb Res. 2020 Jan;185:135-141. doi: 10.1016/j.thromres.2019.11.010. Epub 2019 Nov 13. PMID 31816553
- [Background] Kim BJ, Kwon SU, Park JM, Hwang YH, Heo SH, Rha JH, Lee J, Park MS, Kim JT, Song HJ, Park JH, Yu S, Lee SJ, Park TH, Cha JK, Kwon HM, Kim EG, Lee SH, Lee JS, Lee J, Kang DW. Blood Pressure Variability Is Associated With White Matter Lesion Growth in Intracranial Atherosclerosis. Am J Hypertens. 2019 Aug 14;32(9):918-924. doi: 10.1093/ajh/hpz068. PMID 31044227